CLINICAL TRIAL: NCT06816095
Title: Gene and Molecular Pathway Characterization of the Response to Ozone Treatment in Gynecological Tumor Patients With Chronic Pelvic Pain Secondary to Radio-chemotherapy
Brief Title: Gene and Molecular Pathways of Ozone Treatment Response in Gynecological Tumor Patients With Chronic Pelvic Pain Secondary to Cancer Treatment
Acronym: OzoGynEpigen
Status: Recruiting | Type: Observational
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other); Fundación DISA, Canary Islands, Spain (Unknown); Council of Gran Canaria (Other)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, Head of the Research Unit, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: 2024-192-1; DISA'24: OA24/104 (Other Grant/Funding Number: Fundación DISA); CIGC'23/24 (Other Grant/Funding Number: Cabildo de Gran Canaria)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pelvic Pain Syndrome (CPPS); Radiation-Induced Disorder; Radiotherapy Side Effects; Side Effect of Chemotherapy; Gynecological Cancers
Keywords: Radiation-Induced Disorder; Radiotherapy Side Effects; Cancer survivors; Chronic Pelvic Pain Syndrome (CPPS); Gynecological Cancers; gene expression; epigenetic clocks; side effects of cancer treatment; Toxicity of chemotherapy; Ozone therapy; Quality of Life; oxidative stress
MeSH Terms: conditions — Abnormalities, Radiation-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treated patients, without secondary pain: Patients with gynecological tumors, treated with radiotherapy/chemotherapy, without chronic pelvic pain.
- Treated patients, with chronic pelvic pain: Patients with gynecological tumors, treated with radiotherapy/chemotherapy, with chronic pelvic pain, submitted to our Chronic Pain Unit for compassionate/palliative ozone treatment.

SUMMARY:
Gynecological cancers, including those affecting the ovaries, uterus, and cervix, represent a significant health burden for women. While survival rates have improved, many women experience chronic pelvic pain secondary to cancer treatment, especially radiotherapy and chemotherapy. This treatment-induced pelvic pain can be of difficult management and significantly affects patients' quality of life.

In our experience, ozone therapy has emerged as a promising complementary treatment for pain relief in patients with chronic diseases, including side effects of cancer treatment. However, the genetic and epigenetic mechanisms influencing its effectiveness have not yet been thoroughly studied.

The aim of this prospective study is to analyze how ozone therapy modulates the expression of certain genes and its impact on epigenetic clocks, which could help predict pain response.

DETAILED DESCRIPTION:
While survival rates of gynecological cancers have improved, many women experience chronic pelvic pain as a consequence of cancer treatment, particularly radiotherapy and chemotherapy. This persistent pain often has neuropathic characteristics, and it can be challenging to manage, negatively impacting physical and emotional well-being and quality of life.

Conventional pain management strategies for these patients often provide limited relief. In our experience, ozone therapy has emerged as a promising option for managing chronic pain in various conditions, including side effects of cancer treatment.

While the clinical benefits of ozone therapy have been observed in preliminary studies, the underlying molecular mechanisms underlying its analgesic effect remain largely unknown. Understanding how ozone therapy influences gene expression and epigenetic modifications could facilitate the identification of genes involved in the differential response to ozone therapy and a potential way for personalized strategies for pain treatment.

The aim of this prospective study is to analyze how ozone therapy modulates the expression of certain genes and its impact on epigenetic clocks, which could help predict pain response.

Primary Objectives:

In patients with gynecological tumors treated by radiotherapy/chemotherapy, To evaluate

* among patients with or without chronic pelvic pain induced by treatment.
* before and after ozone treatment in those patients treated because of pelvic pain induced by radiotherapy/chemotherapy.

The potential differences in:

1. Gene expression.
2. Biological age based on epigenetic clocks:

Secondary Objectives:

Evaluate in those patients the potential relationship between gene expression and epigenetic clocks with:

1. Grade of toxicity
2. Pain score
3. Health-related quality of life,
4. Biochemical markers of oxidative stress and inflammation.

Trial Design:

This observational and prospective study will analyze data from two groups of patients with gynecological tumors treated with radiotherapy/chemotherapy:

* A group of patients with chronic pelvic pain secondary to radiotherapy-chemotherapy, submitted to our Chronic Pain Unit for compassionate/palliative ozone treatment.
* A group of patients without secondary chronic pelvic pain.

Trial Population:

Adult women (≥ 18 years old) with gynecological tumors treated with radiotherapy-chemotherapy. They will be analyzed into two different groups of patients:

* A group of patients with chronic pelvic pain secondary to radiotherapy-chemotherapy, submitted to our Chronic Pain Unit for compassionate/palliative ozone treatment.
* A group of patients without secondary chronic pelvic pain.

Intervention. No intervention. The management of patients will be the standard of care in our hospital.

Study Duration:

The primary completion date is planned for 14/February/2027. The study completion date is planned for 14/August/2027

ELIGIBILITY:
Inclusion Criteria:

* Adult women (>=18 years old) with gynecological tumors treated with radiotherapy-chemotherapy.
* Cancer disease is stable or in remission.
* Life expectancy > = 6 months.
* Patients included in the group of patients with pelvic pain must have a clinical, radiological, endoscopic, or histopathological diagnosis that their pain is not secondary to the oncological process.
* Patients included in the group of patients with pelvic pain must have pain for >= 3 months duration, with an intensity >= 3 on the Visual Analog Scale (VAS), or classified as toxicity >= Grade-2 of the CTCAE v.5.0 of the National Cancer Institute of the USA.
* Signed and dated informed consent specific to this study.

Exclusion Criteria:

* Age < 18 years old.
* Severe psychiatric disorders.
* Inability to complete the quality of life questionnaires.
* Active neoplasia requiring recent initiation (< 3 months) of systemic or local treatment.
* Life expectancy (for any reason) < 6 months.
* Failure to meet all inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women with female reproductive organs who are at risk for gynecological cancers
Study Population: Adult women (≥18 years) with gynecological tumors treated with radiotherapy-chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-02-14 (Estimated); Study Completion 2027-08-14 (Estimated)

PRIMARY OUTCOMES:
Differences in gene expression among patients with or without chronic pelvic pain induced by radiotherapy/chemotherapy. | At 0 week
  Differences (among patients with or without chronic pelvic pain induced by radiotherapy/chemotherapy) in gene expression profile.
Changes (from baseline) in gene expression at the end of ozone treatment. | At 16 weeks
  Changes (from baseline) in gene expression profile, after ozone treatment.
Differences in biological age based on epigenetic clocks among patients with or without chronic pelvic pain induced by radiotherapy/chemotherapy | At 0 week.
  Differences (among patients with or without chronic pain induced by radiotherapy/chemotherapy) in the biological age based on epigenetic clocks.
Changes (from baseline) in the biological age based on epigenetic clocks, after ozone treatment | At 16 weeks.
  Changes (from baseline) in the biological age based on epigenetic clocks, after ozone treatment

SECONDARY OUTCOMES:
Differences in the grade of toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 scale among patients with or without chronic pain induced by radiotherapy/chemotherapy | At 0 week.
  Differences (among patients with or without chronic pain induced by radiotherapy/chemotherapy) in the grade of toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 scale (from the National Cancer Institute of EEUU). Range from: Grade = (asymptomatic or mild symptoms) to Grade 3 (severe symptoms, limiting self-care activities in daily life).
Changes (from baseline) in the grade of toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 scale, after ozone treatment. | At 16 weeks.
  Changes (from baseline) in the grade of toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 scale (from the National Cancer Institute of EEUU). Range from: Grade = (asymptomatic or mild symptoms) to Grade 3 (severe symptoms, limiting self-care activities in daily life).
Differences in pain score according to the visual analog scale (VAS) among patients with or without chronic pain induced by radiotherapy/chemotherapy | At 0 week.
  Self-reported evaluation of the severity of pain according to the VAS, scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine").
Change (from baseline) in pain score according to the visual analog scale (VAS), after ozone treatment. | At 16 weeks.
  Self-reported evaluation of the severity of pain according to the VAS, scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine").
Differences in "Quality of Life" (using the EQ-5D-5L questionnaire) self-perceived by patients among patients with or without chronic pain induced by radiotherapy/chemotherapy. | At 0 week.
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (Best: I have no problem) to 5 (worst: I have an extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analog scale (0 = worst health patient can imagine, 100 = best health patient can imagine).
Changes (from baseline) in "Quality of Life" (using the EQ-5D-5L questionnaire) self-perceived by patients, after ozone treatment. | At 16 weeks.
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (Best: I have no problem) to 5 (worst: I have an extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analog scale (0 = worst health patient can imagine, 100 = best health patient can imagine).
Differences in biochemical parameters of oxidative stress among patients with or without chronic pain induced by radiotherapy/chemotherapy. | At 0 week.
  Differences in serum levels of antioxidants and free radicals.
Changes (from baseline) in biochemical parameters of oxidative stress, after ozone treatment. | At 16 weeks.
  Changes in serum levels of antioxidants and free radicals.
Differences in biochemical parameters of inflammation among patients with or without chronic pain induced by radiotherapy/chemotherapy. | At 0 week.
  Differences in serum levels of pro-inflammatory cytokines.
Changes (from baseline) in biochemical parameters of inflammation, after ozone treatment. | At 16 weeks.
  Changes in serum levels of pro-inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhD, Study Chair — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain.; Francisco Rodríguez-Esparragón, BSc, PhD, Study Director — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain.; Sara Cazorla-Rivero, BSc, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain.; Mario Federico, MD, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Spain.
Locations (1):
- Hospital Universitario de Gran Canaria Dr. Negrín, (FIISC), Las Palmas, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Yes
It will be available (after request):
  * Individual participant data (IPD) that underlie the results reported in further articles, after deidentification
  * Data will be available after publication, ending 36 months following article publication.
  * They will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  * Study protocol
  Proposals should be directed to: bernardinoclavo@gmail.com To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication, ending 36 months following article publication.
Access Criteria: Data will be available for investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  - Study protocol
  Proposals should be directed to: bernardinoclavo@gmail.com To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Tricarico G, Travagli V. The Relationship between Ozone and Human Blood in the Course of a Well-Controlled, Mild, and Transitory Oxidative Eustress. Antioxidants (Basel). 2021 Dec 4;10(12):1946. doi: 10.3390/antiox10121946. PMID 34943049
- [Background] Hidalgo-Tallon FJ, Torres-Morera LM, Baeza-Noci J, Carrillo-Izquierdo MD, Pinto-Bonilla R. Updated Review on Ozone Therapy in Pain Medicine. Front Physiol. 2022 Feb 23;13:840623. doi: 10.3389/fphys.2022.840623. eCollection 2022. PMID 35283802
- [Background] Galie M, Covi V, Tabaracci G, Malatesta M. The Role of Nrf2 in the Antioxidant Cellular Response to Medical Ozone Exposure. Int J Mol Sci. 2019 Aug 17;20(16):4009. doi: 10.3390/ijms20164009. PMID 31426459
- [Background] Clavo B, Santana-Rodriguez N, Llontop P, Gutierrez D, Ceballos D, Mendez C, Rovira G, Suarez G, Rey-Baltar D, Garcia-Cabrera L, Martinez-Sanchez G, Fiuza D. Ozone Therapy in the Management of Persistent Radiation-Induced Rectal Bleeding in Prostate Cancer Patients. Evid Based Complement Alternat Med. 2015;2015:480369. doi: 10.1155/2015/480369. Epub 2015 Aug 18. PMID 26357522
- [Background] Clavo B, Rodriguez-Esparragon F, Rodriguez-Abreu D, Martinez-Sanchez G, Llontop P, Aguiar-Bujanda D, Fernandez-Perez L, Santana-Rodriguez N. Modulation of Oxidative Stress by Ozone Therapy in the Prevention and Treatment of Chemotherapy-Induced Toxicity: Review and Prospects. Antioxidants (Basel). 2019 Nov 26;8(12):588. doi: 10.3390/antiox8120588. PMID 31779159
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Long-Term Results with Adjuvant Ozone Therapy in the Management of Chronic Pelvic Pain Secondary to Cancer Treatment. Pain Med. 2021 Sep 8;22(9):2138-2141. doi: 10.1093/pm/pnaa459. No abstract available. PMID 33738491
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Ozone Therapy in Refractory Pelvic Pain Syndromes Secondary to Cancer Treatment: A New Approach Warranting Exploration. J Palliat Med. 2021 Jan;24(1):97-102. doi: 10.1089/jpm.2019.0597. Epub 2020 May 5. PMID 32379556
- [Background] Clavo B, Rodriguez-Abreu D, Galvan S, Federico M, Martinez-Sanchez G, Ramallo-Farina Y, Antonelli C, Benitez G, Rey-Baltar D, Jorge IJ, Rodriguez-Esparragon F, Serrano-Aguilar P. Long-term improvement by ozone treatment in chronic pain secondary to chemotherapy-induced peripheral neuropathy: A preliminary report. Front Physiol. 2022 Aug 30;13:935269. doi: 10.3389/fphys.2022.935269. eCollection 2022. PMID 36111149
- [Background] Clavo B, Martinez-Sanchez G, Rodriguez-Esparragon F, Rodriguez-Abreu D, Galvan S, Aguiar-Bujanda D, Diaz-Garrido JA, Canas S, Torres-Mata LB, Fabelo H, Tellez T, Santana-Rodriguez N, Fernandez-Perez L, Marrero-Callico G. Modulation by Ozone Therapy of Oxidative Stress in Chemotherapy-Induced Peripheral Neuropathy: The Background for a Randomized Clinical Trial. Int J Mol Sci. 2021 Mar 10;22(6):2802. doi: 10.3390/ijms22062802. PMID 33802143
- [Background] Clavo B, Canovas-Molina A, Ramallo-Farina Y, Federico M, Rodriguez-Abreu D, Galvan S, Ribeiro I, Marques da Silva SC, Navarro M, Gonzalez-Beltran D, Diaz-Garrido JA, Cazorla-Rivero S, Rodriguez-Esparragon F, Serrano-Aguilar P. Effects of Ozone Treatment on Health-Related Quality of Life and Toxicity Induced by Radiotherapy and Chemotherapy in Symptomatic Cancer Survivors. Int J Environ Res Public Health. 2023 Jan 13;20(2):1479. doi: 10.3390/ijerph20021479. PMID 36674232
- [Background] Clavo B, Canovas-Molina A, Diaz-Garrido JA, Canas S, Ramallo-Farina Y, Laffite H, Federico M, Rodriguez-Abreu D, Galvan S, Garcia-Lourve C, Gonzalez-Beltran D, Carames MA, Hernandez-Fleta JL, Serrano-Aguilar P, Rodriguez-Esparragon F. Effects of ozone therapy on anxiety and depression in patients with refractory symptoms of severe diseases: a pilot study. Front Psychol. 2023 Aug 4;14:1176204. doi: 10.3389/fpsyg.2023.1176204. eCollection 2023. PMID 37599784
- [Background] Clavo B, Rodriguez-Abreu D, Galvan-Ruiz S, Federico M, Canovas-Molina A, Ramallo-Farina Y, Antonilli C, Benitez G, Fabelo H, Garcia-Lourve C, Gonzalez-Beltran D, Jorge IJ, Rodriguez-Esparragon F, Callico GM. Long-Term Effects of Ozone Treatment in Patients with Persistent Numbness and Tingling Secondary to Chemotherapy-Induced Peripheral Neuropathy. A Retrospective Study. Integr Cancer Ther. 2025 Jan-Dec;24:15347354241307038. doi: 10.1177/15347354241307038. PMID 39797612
- [Background] Bocci VA, Zanardi I, Travagli V. Ozone acting on human blood yields a hormetic dose-response relationship. J Transl Med. 2011 May 17;9:66. doi: 10.1186/1479-5876-9-66. PMID 21575276
- [Background] Bocci V, Valacchi G. Nrf2 activation as target to implement therapeutic treatments. Front Chem. 2015 Feb 2;3:4. doi: 10.3389/fchem.2015.00004. eCollection 2015. PMID 25699252
- [Background] Bocci V, Borrelli E, Travagli V, Zanardi I. The ozone paradox: ozone is a strong oxidant as well as a medical drug. Med Res Rev. 2009 Jul;29(4):646-82. doi: 10.1002/med.20150. PMID 19260079